CLINICAL TRIAL: NCT06645418
Title: Relative Hand Grip Strength and Functional Fitness Among Elderly Patients with Type II Diabetes in Egypt: a Cross-sectional Study
Brief Title: Relative Hand Grip Strength and Functional Fitness in Diabetic Patient in Egypt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mohammed Youssef Elhamrawy, Lecturer of Physical therapy, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Hand Grip
Record Dates: First submitted 2024-10-12; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diabetic group (Active Comparator): 100 randomly selected older adults with DM II, of both sexes who are attending endocrine outpatient clinics in governmental hospitals.
  Interventions: Diagnostic Test: relative Hand grip strength; Diagnostic Test: senior fitness test
- non diabetic group (Active Comparator): 100 older adults non diabetic, of both sexes who are attending endocrine outpatient clinics in governmental hospitals.
  Interventions: Diagnostic Test: relative Hand grip strength; Diagnostic Test: senior fitness test

INTERVENTIONS:
Diagnostic Test: relative Hand grip strength — To perform this study the relative handgrip strength (rHGS) index was used. The rHGSi is defined as the sum of the handgrip strength of both hands divided by body mass index (BMI), and it is considered a better prognostic tool than handgrip strength. rHGS was measured by Jamar hand dynamometer. The Functional Performance was determined by using 3 tests of the Senior Fitness Test (The 30-second chair stand test, the 8-feet Up-and-Go test, and the 2 minutes' Walk Test).
Diagnostic Test: senior fitness test — The Functional Performance was determined by using 3 tests of the Senior Fitness Test (The 30-second chair stand test, the 8-feet Up-and-Go test, and the 2 minutes' Walk Test).

SUMMARY:
To show if there is significant relationship between hand grip strength and physical fitness in diabetic type II patients over 60 years old.

DETAILED DESCRIPTION:
To show if there is significant relationship between hand grip strength and physical fitness in diabetic type II patients over 60 years old.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type II
* Ability to walk independently
* The cognitive and mental capacity to understand and perform tests

Exclusion Criteria:

* Musculoskeletal, neurological, rheumatological problems, or hand deformities that could hinder grasping

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-10-05 (Actual); Study Completion 2024-10-05 (Actual)

PRIMARY OUTCOMES:
relative Hand grip strength | Baseline
  the sum of the handgrip strength of both hands divided by body mass index (BMI)
The 30-Second Chair Test | Baseline
  The 30-Second Chair Test is a standing exercise where participants sit in a folding chair without arms, with their feet shoulder-width apart and arms crossed. The test requires the participant to perform full stands within 30 seconds, with the goal of completing the task without using their arms.
8-feet Up-and-Go test | Baseline
  Place a chair and marker 8 feet apart, clear the path, and start seated. Start timing, then quickly stand, walk, and walk around a cone, returning to the chair. Stop timing as needed. Perform two trials.
2 min walk test | Baseline
  For two minutes, the person is urged to walk as quickly as they can while remaining safe and independent, and the distance is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Yo Elhamrawy, Principal Investigator — National institute for Gerontology
Locations (2):
- Egypt (2):
  - Kz hospital, Cairo, Elgharbia
  - Kz Hospital, Cairo

IPD SHARING:
Plan to Share IPD: No